CLINICAL TRIAL: NCT03372096
Title: LC Bead LUMI for Prostatic Artery Embolization: A Pilot Study
Brief Title: LC Bead LUMI for Prostatic Artery Embolization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-2782
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Results first posted 2021-02-05 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: BPH
Keywords: embolization; prostate

STUDY DESIGN:
Intervention Model Description: This will be an open label pilot study with a small population undergoing an intervention to determine initial safety and potential for efficacy as measured by improvement of LUTS and decrease in prostate size
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All patients (Experimental): Patients will receive the Prostatic Artery Embolization procedure.
  Interventions: Device: Prostatic Artery Embolization

INTERVENTIONS:
Device: Prostatic Artery Embolization — LC Bead LUMI is a spherical polyvinyl alcohol embolic particle that incorporates radiopaque moieties. Once a catheter has been fluoroscopically guided into the target vessel, the beads are then injected, causing obstruction at the arteriole level until the desired degree of embolization has occurred.
  Other Names: LC Bead LUMI

SUMMARY:
Purpose: The purpose of this pilot study is to determine preliminary estimates of the parameters related to the distribution of the study endpoints including: International Prostate Symptom Score (IPSS) and quality of life (QoL) score changes, Qmax (maximum urine flow rate) changes, post void residual volume (PVR) changes, percent prostate infarction and presence of non-target embolization.

Participants: 20 adult male subjects with benign hyperplasia will be enrolled in this study.

Procedures (methods): This will be a multisite, open label pilot study with a small population undergoing an investigational intervention (prostatic artery embolization) to determine initial safety and potential for efficacy as measured by improvement of lower urinary tract symptoms (LUTS) and decrease in prostate size.

DETAILED DESCRIPTION:
This will be an open label pilot study with a small population undergoing an intervention to determine initial safety and potential for efficacy as measured by improvement of LUTS and decrease in prostate size

ELIGIBILITY:
Inclusion Criteria

1. Male
2. Age > 40
3. Prostate gland >50 grams as measured by pre-procedural CT angiogram (CTA)
4. Have previously taken BPH medication for 6 months without desired improvement of LUTS or has started medication and stopped due to unwanted side effects
5. Moderate to severe LUTS as defined by IPSS score >18
6. Peak urine flow rate (Qmax) <12 mL/sec
7. Capable of giving informed consent
8. Life expectancy greater than 1 year

Exclusion Criteria

1. Severe vascular disease
2. Uncontrolled diabetes mellitus
3. Immunosuppression
4. Neurogenic bladder and/or sphincter abnormalities secondary to Parkinson's disease, multiple sclerosis, cerebral vascular accident, diabetes, etc.
5. Complete urinary retention
6. Impaired kidney function (serum creatinine level > 1.8 mg/dL or a glomerular filtration rate < 60 as approximated using serum creatinine levels) unless anuric and on dialysis.
7. Confirmed or suspected bladder cancer
8. Urethral strictures, bladder neck contracture, or other potentially confounding bladder pathology
9. Ongoing urogenital infection
10. Previous pelvic radiation or radical pelvic surgery
11. Confirmed or suspected malignancy of the prostate based on digital rectal exam (DRE), transrectal ultrasonography (TRUS) or prostate-specific antigen (PSA) (> 10 ng/mL or > 4.0 ng/mL and < 10 ng/mL with free PSA < 25% of total PSA without a negative biopsy).
12. Uncorrectable coagulopathy including international normalized ratio (INR) > 1.5 or platelets < 50,000
13. Contrast hypersensitivity refractory to standard medications (antihistamines, steroids)

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender is based on the anatomical gender assigned at birth. Patients must have a prostate in order to enroll in this study.
Enrollment: 18 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ari Isaacson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - UNC Hospitals, Chapel Hill, North Carolina
  - Vascular Institute of Virginia, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 18
Received Intervention | 10
Completed | 10
Not Completed | 8
Not completed — Study Closed | 8

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
IPSS [Mean (Standard Deviation); unit: units on a scale] — The International Prostate Symptom Score (IPSS) is an 8 item Likert questionnaire (7 symptom questions + 1 quality of life question) with scores ranging from 0 to 5, where 0 is less severe. IPSS is a written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). Total scores are determined to be Mild (1-7), Moderate (8-19), or Severe (20-35).
  units on a scale | 22.5 (4.2)
IIEF [Mean (Standard Deviation); unit: units on a scale] — The International Index of Erectile Function is a 15 question tool that measures erectile function (30 max), orgasmic function (10max), sexual desire (10 max), intercourse satisfaction (15 max), and overall satisfaction (10 max). The total maximum score is 75. Higher scores indicated higher levels of sexual function.
  units on a scale | 46 (22)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The QoL question is a single question included with the IPSS related to the symptoms of the disease benign prostatic hyperplasia (BPH). Lower scores indicate a higher quality of life. The range of this scale is 0 to 5.
  units on a scale | 4.5 (0.7)
Urine Flow (mL/s) [Mean (Standard Deviation); unit: mL/s] — Urine flow will be measured to determine the maximum rate of urine flow (Qmax), which is measured in mL per second. Population: 3 participants never underwent baseline urodynamic testing because they withdrew from the study.
  mL/s
    number analyzed (Participants) | 15
    (all) | 7.9 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in IPSS Score
Description: The International Prostate Symptom Score (IPSS) is an 8 item Likert questionnaire (7 symptom questions + 1 quality of life question) with scores ranging from 0 to 5, where 0 is less severe. IPSS is a written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). Total scores are determined to be Mild (1-7), Moderate (8-19), or Severe (20-35).
Time Frame: Baseline and 6 months following PAE procedure
Population: This group includes all subjects that received the PAE procedure with 6 month follow up IPSS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients With 6 Month Follow up: Patients will receive the Prostatic Artery Embolization procedure.
  Prostatic Artery Embolization: LC Bead LUMI is a spherical polyvinyl alcohol embolic particle that incorporates radiopaque moieties. Once a catheter has been fluoroscopically guided into the target vessel, the beads are then injected, causing obstruction at the arteriole level until the desired degree of embolization has occurred.
Arm/Group | Patients With 6 Month Follow up
Number analyzed (Participants) | 7
units on a scale | -11.4 (8.4)

2. Secondary Outcome: Mean Change in Quality of Life Scores
Description: The QoL question is a single question included with the IPSS related to the symptoms of the disease benign prostatic hyperplasia (BPH). Lower scores indicate a higher quality of life. The range of this scale is 0 to 5.
Time Frame: Baseline and 6 months following PAE procedure
Population: This group includes all patients that received the PAE procedure and had 6 month QoL data collected.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Patients With 6 Month Follow up Data: Patients will receive the Prostatic Artery Embolization procedure.
  Prostatic Artery Embolization: LC Bead LUMI is a spherical polyvinyl alcohol embolic particle that incorporates radiopaque moieties. Once a catheter has been fluoroscopically guided into the target vessel, the beads are then injected, causing obstruction at the arteriole level until the desired degree of embolization has occurred.
Arm/Group | Patients With 6 Month Follow up Data
Number analyzed (Participants) | 7
units on a scale | -2 (1.3)

3. Secondary Outcome: Mean Change in Urine Flow
Description: Urine flow will be measured to determine the maximum rate of urine flow (Qmax), which is measured in mL per second.
Time Frame: Baseline and 6 months following PAE Procedure
Population: Patients with 6-month urodynamic testing
Measure: Mean (Standard Deviation); unit: mL/s
Groups:
- All Patients With 6 Month Uroflow Testing: Patients will receive the Prostatic Artery Embolization procedure.
  Prostatic Artery Embolization: LC Bead LUMI is a spherical polyvinyl alcohol embolic particle that incorporates radiopaque moieties. Once a catheter has been fluoroscopically guided into the target vessel, the beads are then injected, causing obstruction at the arteriole level until the desired degree of embolization has occurred.
Arm/Group | All Patients With 6 Month Uroflow Testing
Number analyzed (Participants) | 6
mL/s | 3.3 (4.5)

4. Secondary Outcome: Mean Change in Prostate Volume
Description: Change in the prostate volume measured in grams.
Time Frame: Baseline and 3 months following
Population: All participants receiving the PAE procedure with imaging following the procedure.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | All Patients
Number analyzed (Participants) | 10
grams | -20 (23.2)

5. Secondary Outcome: Percent of Prostate Infarcted
Description: Percentage of prostate infarcted will be determined using manual demarcation of non-enhancing areas within the prostate on serial axial slices of post contrast CT images. Segmentation software will then be employed to calculate the volume.
Time Frame: 6 months following PAE procedure
Population: Unable to collect infarction data because the CT scans did not show it effectively.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants That Have Non-Targeted Embolization Following the Prostatic Artery Embolization (PAE) Procedure
Description: Number of participants that have non-targeted embolization following the prostatic artery embolization (PAE) procedure. Non-target embolization will be determined by comparing non-contrast CT images from pre- and post-PAE scans or clinical symptoms. This will be a binary data point and not a calculation.
Time Frame: 3 months following PAE procedure
Population: All patients that received the PAE procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 10
Participants | 8

7. Secondary Outcome: Number of Participants That Have Minor Complications Following the Prostatic Artery Embolization (PAE) Procedure
Description: Number of participants that experience minor complications following the PAE procedure.
Time Frame: Up to 12 months following PAE procedure
Population: All patients that received the PAE procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 10
Participants | 8

8. Secondary Outcome: Mean Change in IIEF Score
Description: Change in sexual function as determined by an unchanged or improved score on the International Index of Erectile Function (IIEF) questionnaire. The International Index of Erectile Function is a 15 question tool that measures erectile function (30 max), orgasmic function (10 max), sexual desire (10 max), intercourse satisfaction (15 max), and overall satisfaction (10 max). The total maximum score is 75. Higher scores indicated higher levels of sexual function.
Time Frame: Baseline and 6 months following PAE procedure
Population: All patients that received the PAE procedure and had 6 month follow up data for IIEF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 7
units on a scale | -1.1 (13.4)

ADVERSE EVENTS:
Time Frame: 1 year following PAE procedure
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=10)
brief penile pain and sensitivity (Renal and urinary disorders) | 3 (3)
brief rectalgia or anal pain (Renal and urinary disorders) | 2 (2)
dysuria (Renal and urinary disorders) | 2 (2)
increased frequency (Renal and urinary disorders) | 1 (1)
penile ulceration (Renal and urinary disorders) | 1 (1)
temporary increased urgency to urinate (Renal and urinary disorders) | 2 (2)
temporary hematuria (Renal and urinary disorders) | 1 (1)
temporary urinary retention (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT03372096/Prot_SAP_000.pdf